CLINICAL TRIAL: NCT02116062
Title: Robotic Microsurgery of the Ocular surfaceProspective Human Feasibility Study
Brief Title: Robotic Surgery of the Ocular Surface
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The results concerning amniotic membrane transplantation (n=7) and robot-assisted pterygium surgery (n=5) were conclusive
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5540
Record Dates: First submitted 2014-02-24; First posted 2014-04-16 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Keratitis; Pterygium; Corneal Opacity Corneal Thinning; Corneal Perforation
MeSH Terms: conditions — Keratitis; Pterygium; Corneal Perforation | interventions — Inlays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amniotic membrane transplantation (Other)
  Interventions: Device: 1. Amniotic membrane transplantation on the cornea with the Da Vinci Si HD© robot (Inlay or overlay technique)
- Pterygium surgery (Other)
  Interventions: Device: Pterygium removal and autograft of the conjunctiva with the Da Vinci Si HD© robot (Kenyon technique)
- Penetrating keratoplasty (Other)
  Interventions: Device: Penetrating keratoplasty using Baron trephine and nylon stitches with the Da Vinci Si HD© robot

INTERVENTIONS:
Device: 1. Amniotic membrane transplantation on the cornea with the Da Vinci Si HD© robot (Inlay or overlay technique)
  Arms: Amniotic membrane transplantation
Device: Pterygium removal and autograft of the conjunctiva with the Da Vinci Si HD© robot (Kenyon technique)
  Arms: Pterygium surgery
Device: Penetrating keratoplasty using Baron trephine and nylon stitches with the Da Vinci Si HD© robot
  Arms: Penetrating keratoplasty

SUMMARY:
The introduction of surgical robots in the OR revolutionized a number of specialties (i. e. urology, gynecology, digestive surgery). Robots are currently used in many situations and the list of appropriate indications is growing rapidly. There are many potential advantages of robotics in eye surgery such as increased precision and maneuverability, better ergonomics, improved patient access to surgeons and surgical training. As a result, robotics might improve patient care. The Da Vinci© robot has been used for 10 years in experimental conditions to suture corneal lacerations, to perform corneal grafts, to remove ocular foreign bodies, lens capsules and vitreous. The authors reported a lack of precision resulting from poor visualization and the absence of microsurgical instruments. These elements were considered to be hurdles to further clinical investigation. The new Da Vinci Si HD© robot has been available since 2009 at the IRCAD center and more recently in Strasbourg University Hospital. It provides greater magnification and better resolution of the operative field than the previous model. We performed since 2012 various ocular surface surgeries on porcine eyes at the IRCAD center. The aim of the present trial is to perform the same procedures (amniotic membrane transplantations, pterygium surgeries, corneal grafts) in a clinical setting with the Da Vinci Si HD© system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 18 year-old suffering :

symptomatic pterygium

* chronic corneal ulceration resistant to medical treatment
* corneal opacity involving corneal stroma and corneal endothelium
* corneal thinning
* corneal perforation

Exclusion Criteria:

* History of eye surgery
* psychiatric disease
* mental deficiency
* pregnancy
* nursing mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Respect for different phases of the operating procedure of each intervention. | At the end of the surgery
  Surgeons will check that all steps of the surgery have been done and successfully completed (thanks to a surgery ckeck-list procedure and video tape)

CONTACTS AND LOCATIONS:
Overall Officials: Bourcier Tristan, PHMD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Bourcier T, Chammas J, Becmeur PH, Danan J, Sauer A, Gaucher D, Liverneaux P, Mutter D. Robotically Assisted Pterygium Surgery: First Human Case. Cornea. 2015 Oct;34(10):1329-30. doi: 10.1097/ICO.0000000000000561. PMID 26203760